CLINICAL TRIAL: NCT04027621
Title: Safety and Effectiveness of Remote Ischemic Conditioning Combined With Intravenous Thrombolysis in Treating Acute Ischemic Stroke
Acronym: SERICT-AIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SERICT-AIS
Record Dates: First submitted 2019-07-14; First posted 2019-07-22 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Active Comparator): RIC+Standard medical treatment Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg. RIC will be conducted twice within 6 to 24 hours from thrombolysis. Additionally,the patients will be treated with standard medical treatment according to Guidelines for diagnosis and treatment of acute ischemic stroke in China 2014.
  Interventions: Device: remote ischemic conditioning
- control group (Placebo Comparator): Sham RIC+Standard medical treatment Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg. RIC will be conducted twice twice within 6 to 24 hours from thrombolysis. Additionally,the patients will be treated with standard medical treatment according to Guidelines for diagnosis and treatment of acute ischemic stroke in China 2014
  Interventions: Device: sham remote ischemic conditioning

INTERVENTIONS:
Device: remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg.
  Arms: RIC group
Device: sham remote ischemic conditioning — Sham remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min re-perfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg.
  Arms: control group

SUMMARY:
The purpose of this study is to determine the efficacy and safety of remote ischemic conditioning combined with intravenous thrombolysis in treating acute ischemic stroke.

DETAILED DESCRIPTION:
In this study, cases of ischemic stroke who undergo intravenous thrombolysis within 4.5 hours from onset are included. The experimental group receive basic treatment and remote ischemic conditioning for 200mmHg, 2 times within 6 hours to 24 hours from thrombolysis. The control group receive basic treatment and remote ischemic conditioning control for 60mmHg, 2 times within 6 hours to 24 hours from thrombolysis . Two groups will be followed up for 90 days to evaluate the efficacy and safety of remote ischemic conditioning combined with intravenous thrombolysis in treating acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age≥18 years, < 80 years, regardless of sex;
* 2) Patients with clinically definite diagnosis of acute ischemic stroke and undergo intravenous thrombolysis;
* 3) Baseline NIHSS >= 5, and <= 25;
* 4) Baseline GCS ≥8;
* 5) Signed and dated informed consent is obtained

Exclusion Criteria:

* 1) Patients who undergo endovascular treatment;
* 2) mRS ≥ 2 before the onset of the disease;
* 3) Double upper limbs or lower limbs paralysis was found in this case;
* 4) Active bleeding of organs within 6 months of admission or current, including cerebral hemorrhage, subarachnoid hemorrhage, gastrointestinal hemorrhage, fundus hemorrhage and so on;
* 5) Other intracranial lesions, such as cerebrovascular malformation cerebral venous diseases, tumor and other diseases involving the brain;
* 6) Concurrent use of anticoagulation drugs including Warfarin, dabigatran, rivaroxaban;
* 7) Severe organ dysfunction or failure;
* 8) Patients suffering from severe hematological diseases or severe coagulation disorder dysfunction
* 9) Those who have a history of severe trauma or had major surgery within 6 months prior to admission;
* 10) Those who have a history of atrial fibrillation;
* 11) The patients who have the contraindication of remote ischemic conditioning treatment, such as severe soft tissue injury, fracture or vascular injury in the upper limb#Acute or subacute venous thrombosis, arterial occlusive disease, subclavian steal syndrome, etc;
* 12) Pregnant or lactating women;
* 13) Previous remote ischemic conditioning therapy or similar treatment;
* 14) Patients with a life expectancy of less than 3 months or patients unable to complete the study for other reasons;
* 15) Severe hepatic and renal dysfunction;
* 16) Unwilling to be followed up or treated for poor compliance;
* 17) He/She is participating in other clinical research or has participated in other clinical research or has participated in this study within 3 months prior to admission;
* 18) Other conditions that the researchers think are not suitable for the group.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events during hospitalization | 7 days
  All adverse events until day-7 or discharge (whichever is earlier)
Frequency of adverse events during follow-up | 3 months
  Severe adverse events through day-90 after the onset of acute ischemic stroke.

SECONDARY OUTCOMES:
National Institute of Health stroke scale (NIHSS) at 7 days from onset or discharge | 7 days
  National Institute of Health stroke scale (NIHSS) at 7 days from onset or discharge. Ranged from 0 to 42, a low value represents a better outcome.
Proportion of patients with Modified Rankin Scale (mRS) Score 0-2 | 3 months
  Proportion of patients with Modified Rankin Scale (mRS) Score 0-2. Ranged from 0 to 6, a low value represents a better outcome.

OTHER OUTCOMES:
Changes of hematological indicators | 24 hours
  Hematological samples are collected at right before thrombolysis and 24 hours after thrombolysis, and changes of hematological indicators related to hemorrhagic transformation (such as Axl, ANGPTL4) are compared between the two groups.
Changes of the function of dynamic cerebral autoregulation | 10 days
  The function of patients' dynamic cerebral autoregulation are tested 3 times within 10 days from onset and compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China